CLINICAL TRIAL: NCT00320632
Title: Psychopharmacology of Biogenic Amines in Depression
Brief Title: Desipramine for Improving Cellular Signaling and Decreasing Symptoms of Major Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Harvard Medical School (HMS and HSDM) (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, JohnMooney, Principal Investigator, Harvard Medical School (HMS and HSDM)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R01MH015413 (NIH); R01MH015413 (NIH)
Record Dates: First submitted 2006-04-28; First posted 2006-05-03 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2015-08

CONDITIONS: Depression
Keywords: Major Depressive Disorder; MDD
MeSH Terms: conditions — Depression; Depressive Disorder, Major | interventions — Desipramine

INTERVENTIONS:
Drug: Desipramine

SUMMARY:
This study will determine the effectiveness of desipramine in improving cellular signaling, and thereby decreasing symptoms of depression in people with major depressive disorder (MDD).

DETAILED DESCRIPTION:
MDD is a serious mental illness that can interfere with a person's ability to eat, sleep, work, and enjoy activities that were once pleasurable. It is characterized by several symptoms, including as the following: persistent sad, anxious, or "empty" mood; feelings of hopelessness or pessimism; and feelings of guilt, worthlessness, or helplessness. The receptor-G protein-adenylate cyclase enzyme complex (AC enzyme complex) is a major cell signaling system in the brain, blood, and other tissues in the body. Changes in this signaling system among blood cells have been observed in people with major depressive disorder. Research has shown that treatment with the benzodiazepine alprazolam corrects the signaling problem, and thereby improves symptoms of MDD. This study will determine whether impairments in the AC enzyme complex exist among depressed individuals. This study will also evaluate the effectiveness of desipramine, an antidepressant, in improving blood cell signaling, and thereby decreasing symptoms of depression in people with major depressive disorder.

Both healthy and depressed participants will be recruited for this study. All depressed participants in this study will first be assessed for depression severity using the Hamilton Depression Rating Scale. If eligible for the study, participants will be examined to determine AC enzyme complex functioning in both platelets and mononuclear leukocytes. A cohort of the depressed participants will be treated with desipramine. They will be examined to determine the drug's effect on AC enzyme complex functioning, as well as its effect on MDD symptoms, at Weeks 1, 4, and 6.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of MDD (as defined by SCID [DSM III-R] and a score of at least 15 on the 21-item Hamilton Depression Scale)
* Able to swallow tablets, give urine and blood samples, and participate in periodic evaluations during the study
* Healthy volunteers show no current Axis I or Axis II disorders and score less than 8 on the Hamilton Depression Scale

Exclusion Criteria:

* Use of any of the following medications within the 2 weeks prior to study entry: psychoactive medication; aspirin; or nonsteroidal anti-inflammatory agents
* Any alcohol or drug abuse within the 6 months prior to study entry
* Any major medical disorder

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43
Dates: Start 1990-08; Study Completion 1993-07

PRIMARY OUTCOMES:
Measured at Weeks 1, 4, and 6: Catecholamine metabolism and blood cell adenylate cyclase activity
Score on the 21-item Hamilton Depression Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J. Schildkraut, MD, Principal Investigator — Department of Psychiatry, Harvard Medical School
Locations (1):
- Massachusetts Mental Health Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Mooney JJ, Schatzberg AF, Cole JO, Kizuka PP, Salomon M, Lerbinger J, Pappalardo KM, Gerson B, Schildkraut JJ. Rapid antidepressant response to alprazolam in depressed patients with high catecholamine output and heterologous desensitization of platelet adenylate cyclase. Biol Psychiatry. 1988 Mar 15;23(6):543-59. doi: 10.1016/0006-3223(88)90002-9. PMID 2833319
- [Background] Mooney JJ, Samson JA, McHale NL, Colodzin R, Alpert J, Koutsos M, Schildkraut JJ. Signal transduction by platelet adenylate cyclase: alterations in depressed patients may reflect impairment in the coordinated integration of cellular signals (coincidence detection). Biol Psychiatry. 1998 Apr 15;43(8):574-83. doi: 10.1016/s0006-3223(97)00327-2. PMID 9564442
- [Derived] Mooney JJ, Samson JA, Hennen J, Pappalardo K, McHale N, Alpert J, Koutsos M, Schildkraut JJ. Enhanced norepinephrine output during long-term desipramine treatment: a possible role for the extraneuronal monoamine transporter (SLC22A3). J Psychiatr Res. 2008 Jul;42(8):605-11. doi: 10.1016/j.jpsychires.2007.07.009. Epub 2007 Aug 28. PMID 17727882